CLINICAL TRIAL: NCT05377658
Title: A Single-Arm, Phase II Study of AK104 With Chemotherapy as Neoadjuvant and Adjuvant Therapy for Resectable Non-small Cell Lung Cancer
Brief Title: AK104 With Chemotherapy as Neoadjuvant and Adjuvant Therapy for Resectable Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Huijuan Wang, chief physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-005
Record Dates: First submitted 2022-05-10; First posted 2022-05-17 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: neoadjuvant and adjuvant therapy; bispecific antibody
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104+albumin-bound paclitaxel+carboplatin (Experimental): Participants receive 3 cycles of AK104 in combination with albumin-bound paclitaxel and carboplatin as neoadjuvant therapy prior to surgery; followed by surgery; followed by adjuvant AK104 for 9 cycles.
  Interventions: Drug: AK104; Drug: Albumin-Bound Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: AK104 — 10 mg/kg via intravenous infusion on Day 1 of each 21-day cycle.
  Other Names: Cadonilimab
Drug: Albumin-Bound Paclitaxel — 260mg/m^2 via intravenous infusion on Day 1 of each 21-day cycle.
Drug: Carboplatin — AUC 5 mg/mL/min via intravenous infusion on Day 1 of each 21-day cycle.

SUMMARY:
AK104, a tetravalent bispecific antibody targeting PD-1 and CTLA-4, is designed to retain the efficacy benefit of combination of PD-1 and CTLA-4 and improve on the safety profile of the combination therapy. The aim of this study is to evaluate the efficacy and safety of AK104 with chemotherapy as neoadjuvant and adjuvant therapy for patients with resectable stage II-IIIA NSCLC.

ELIGIBILITY:
Key Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
2. Have previously untreated and pathologically confirmed resectable Stage II-IIIA NSCLC.
3. Have at least one measurable lesion per RECIST 1.1 assessed by investigator.
4. Have adequate organ function.

Key Exclusion Criteria:

1. Mixed NSCLC and small cell lung cancer histology.
2. Patients with other active malignancies within 3 years prior to enrollment.
3. Known active autoimmune diseases.
4. Use of immunosuppressive agents within 14 days prior to the first dose of study treatment.
5. Presence of other uncontrolled serious medical conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate | At time of surgery
  defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.

SECONDARY OUTCOMES:
Major Pathological Response (MPR) Rate | At time of surgery
  defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes following completion of neoadjuvant therapy.
Incidence of Surgical Complications | Up to approximately 30 days following surgery
  defined as ≥ grade 3 or severe intraoperative and perioperative complications.
Complete (R0) Resection Rate | After surgery (approximately 7 weeks)
  defined as the percentage of participants achieving complete surgical resection following completion of neoadjuvant therapy.
Objective Response Rate (ORR) | At the end of 3 cycles of neoadjuvant therapy (each cycle is 21 days)
  defined as the percentage of participants having complete response or partial response to protocol treatment. Objective response will be measured by RECIST 1.1.
Event Free Survival (EFS) | Up to approximately 5 years
  defined as the time from the first dose of study drug to disease progression per RECIST 1.1 that precludes surgery, local or distant recurrence, or death due to any cause, whichever occurs first.
Adverse Events (AEs) | From the first dose of neoadjuvant treatment until 90 days after the last dose of adjuvant treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China